CLINICAL TRIAL: NCT05104515
Title: A Phase 1, Multicentre, Open-label, Nonrandomised, First-in-human Study of OVM-200 as a Therapeutic Vaccine in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer, Ovarian Cancer, and Prostate Cancer
Brief Title: First-in-human Study of OVM-200 as a Therapeutic Cancer Vaccine
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oxford Vacmedix UK Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OVM-200-100
Record Dates: First submitted 2021-09-29; First posted 2021-11-03 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer; Non Small Cell Lung Cancer; Ovarian Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: The first part (Phase 1a) comprises a first-in-human (FIH) multiple-dose, sequential-cohort 3+3 design to establish a dose of OVM-200 that is safe and tolerable, and that elicits an immune response in humans.
  This dose will be taken forward into the second part (Phase 1b) of the study. Phase 1b will further assess the safety and tolerability of the selected dose and investigate the immune and tumour response in 3 expansion cohorts of additional patients with NSCLC, ovarian cancer, and prostate cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OVM-200 (Experimental): 2 mg/mL OVM-200 solution. Proposed dose levels for Phase 1a: 250, 500, and 1000 μg. The planned doses may be adjusted based on SRC recommendations. Following review of the data, 1 additional dose level may be added up to a maximum of 2000 μg.
  The dose level for Phase 1b will be selected following review of the data from Phase 1a and will not exceed the dose safely administered in Phase 1a.
  Interventions: Biological: OVM-200

INTERVENTIONS:
Biological: OVM-200 — The first part (Phase 1a) comprises a first-in-human (FIH) multiple-dose, sequential-cohort 3+3 design to establish a dose of OVM-200 that is safe and tolerable, and that elicits an immune response in humans.
  This dose will be taken forward into the second part (Phase 1b) of the study. Phase 1b will further assess the safety and tolerability of the selected dose and investigate the immune and tumour response in 3 expansion cohorts of additional patients with NSCLC, ovarian cancer, and prostate cancer.

SUMMARY:
OVM-200 will be tested in humans for the first time in Study OVM-200-100. Up to 52 patients aged 18-75 with prostate, lung or ovarian cancer will be enrolled in the Study to find out if OVM-200 is safe to continue studying it in patients with cancer. The Study consists of 2 parts: a dose escalation part and a dose expansion part. In the dose escalation part, up to 4 increasing doses of OVM-200 will be evaluated in small groups of cancer patients to find the recommended dose for the expansion part. The recommended dose of OVM-200 will then be given to cancer patients in the dose expansion part to confirm safety and understand how effective it is against their disease and if there are any side effects.

Patients who agree to participate in the Study and pass screening will receive 3 doses of OVM-200 in total at 2-week intervals as an injection under the skin. After completing treatment with OVM-200 patients will be followed up for side effects and to monitor changes in their cancer. Patients will stay on the Study for about 6 months in total during which they will have 10 hospital visits. The Study will run at around 5 sites in the UK.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed metastatic or locally advanced inoperable NSCLC, ovarian cancer, or prostate cancer that have already received at least 1 line of approved cancer therapy and either: exhausted current recognized treatment options; or are stable in a planned treatment-free interval following completion of a set course of treatment; or in the case of prostate cancer, are currently stable on an antihormonal treatment.

  2. Are not receiving active cancer treatment other than supportive therapies or androgen deprivation therapies for prostate cancer, which may be continued, and, in the opinion of the investigator, are not anticipated to require further approved cancer treatment options until the Week 8 assessment (up to 9 weeks) after the first dose of OVM-200 per standard of care.

  3. At least 1 measurable lesion that can be accurately assessed at baseline by computed tomography (CT)/magnetic resonance imaging (MRI) and is suitable for repeated assessment (NSCLC only).

  4. Age ≥ 18 years and ≤ 75 years. 5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Section 7.2.6).

  6. Predicted life expectancy ≥ 3 months. 7. Adequate bone marrow, renal, and hepatic function.

Exclusion Criteria:

1. Known history or evidence of significant immunodeficiency due to underlying illness. Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisolone equivalent) or other immunosuppressive medications within 14 days of the first dose of study drug. Inhaled or topical steroids and adrenal replacement steroids are permitted in the absence of autoimmune disease.
2. Patients with a history of or active, known, or suspected autoimmune disease or a syndrome that requires systemic or immunosuppressive agents. Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune disease only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enrol.
3. Prior therapy with an anticancer vaccine; anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody; or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways in the 28 days before the first dose of study drug.
4. Administration of an investigational drug in the 28 days or 6 half-lives (whichever is longer) before the first dose of study drug.
5. Major surgery or treatment with any chemotherapy, or radiation therapy for cancer in the 28 days before the first dose of study drug.
6. Active infection requiring antibiotics or physician monitoring, or recurrent fevers (> 38.0°C) associated with a clinical diagnosis of active infection.
7. Active viral disease, positive test for hepatitis B virus using hepatitis B surface antigen test, or positive test for hepatitis C virus (HCV) using HCV ribonucleic acid or HCV antibody test indicating acute or chronic infection. Positive test for human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome; testing is not required in the absence of history.
8. Receipt of any vaccine within 28 days before the first dose of study drug.
9. Other prior malignancy within the previous 3 years, except for local or organ-confined early stage cancer that has been definitively treated with curative intent and does not require ongoing treatment, has no evidence of residual disease, and has a negligible risk of recurrence and is therefore unlikely to interfere with the primary and secondary endpoints of the study, including response rate and safety and tolerability.
10. Symptomatic brain metastases or any leptomeningeal metastasis.
11. Any serious or uncontrolled medical disorder (including cardiovascular, respiratory, renal, or autoimmune disease) that, in the opinion of the investigator or the medical monitor, may increase the risk associated with study participation or study drug administration, impair the ability of the patient to receive protocol therapy, or interfere with the interpretation of study results.
12. History of allergic reaction or hypersensitivity to any component of the OVM-200 therapeutic vaccine or adjuvant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint (safety and tolerability) for this study is the occurrence and intensity of adverse events. | 24 Weeks

SECONDARY OUTCOMES:
Immune response to OVM 200 as measured by ELISpot for T cell responses and ELISA for antibody responses. | 24 Weeks
Disease progression and tumour response evaluated using Response Evaluation Criteria in Solid Tumour (RECIST) | 24 Weeks
In ovarian cancer patients, tumour marker CA-125 measured and evaluated according to Gynecologic Cancer Intergroup Criteria (GCIC). | 24 Weeks
In prostate cancer patients, tumour markers prostate-specific antigen (PSA) and total alkaline phosphatase (ALP) as per PCWG3 response criteria. | 24 Weeks
Survivin expression will be correlated to response (based on immune response, tumour assessments, and tumour marker measurements) achieved after OVM-200 administration. | 24 Weeks

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - University College London Hospitals NHS Foundation Trust, London, London
  - Sarah Cannon Research Institute UK, London
  - The Christie NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wijaya W, Morris T, Forster MD, Flynn M, Tuthill M, Thistlethwaite F, Williams A, Finch W, Lu W, Jiang S. Survivin recombinant overlapping peptide (ROP) vaccine in advanced solid tumours: a first-in-human, multicentre, open-label, phase 1a dose-escalation study. EClinicalMedicine. 2025 Dec 27;91:103717. doi: 10.1016/j.eclinm.2025.103717. eCollection 2026 Jan. PMID 41536940